CLINICAL TRIAL: NCT01865383
Title: Microfinance and Health Intervention Trial for Youth in Dar es Salaam, Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Muhimbili University of Health and Allied Sciences (Other); American University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-1111; 1R01MH098690-01 (NIH)
Record Dates: First submitted 2013-05-24; First posted 2013-05-30 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2017-04

CONDITIONS: Sexually Transmitted Infections; Domestic Violence
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microfinance and Health Leadership (Experimental): Microfinance and Health Leadership: Participants will be eligible to receive small loans and business training as part of the microfinance component. Nominated leaders in camps will receive health leadership training on prevention of HIV risk behaviors and gender based violence perpetration, and then pass on knowledge to camp members.
  Interventions: Behavioral: Microfinance and Health Leadership
- Control (No Intervention): Control: Participants will receive delayed HIV prevention training at the conclusion of the intervention involving participants in the other condition.

INTERVENTIONS:
Behavioral: Microfinance and Health Leadership — Microfinance and Health Leadership: Participants will be eligible to receive small loans and business training as part of the microfinance component. Nominated leaders in camps will receive health leadership training on prevention of HIV risk behaviors and gender based violence perpetration, and then pass on knowledge to camp members.
  Arms: Microfinance and Health Leadership

SUMMARY:
Young men who are members of the camps randomized to receive a microfinance and health leadership intervention will have a lower incidence of sexually transmitted infections (Neisseria gonorrhea (NG), Chlamydia trachomatis (CT) and Trichomonas vaginalis (TV) and report perpetrating less physical or sexual violence against sexual partners as compared to young men who are members of camps not randomized to receive the intervention.

DETAILED DESCRIPTION:
Finding effective strategies to reach out to young men and mobilize them to reduce their HIV risk is critical, given men's control over the terms and conditions of most sexual partnerships. Unequal power distribution in relationships has a devastating impact on women, leading to HIV prevalence among young women in some sub-Saharan African countries four to seven times higher than among young men the same age. Gender power differentials have negative consequences for men as well, leading to increased risk of physical and mental health problems, substance use, and low uptake of health-related services. We need innovative approaches to address the structural and social determinant of young men's risk. Lack of economic opportunity is a key structural determinant of risk that has negative consequences for men, and has been linked to poor health outcomes. The influence of social network members is a social determinant of risk for both HIV and gender-based violence that can be addressed through interventions designed to change network norms. For the past 12 years our group has conducted research in Dar es Salaam, Tanzania on HIV and gender-based violence. With support from the National Institute of Mental Health (NIMH) we identified networks of young men who socialize in what are called "camps" and we successfully piloted a microfinance and health leadership intervention with men in camps like the one proposed in this application (R21 MH080577). Camps are enduring social groups of mostly men that have elected leadership, paid membership fees, and physical space to meet. The equivalent of a camp in US culture may be a cross between a club and a gang. Camps appear to be an urban phenomenon in Tanzania and our group is the first to have published data describing them. Men in camps engage in HIV risk behavior and in gender-based violence that put them and their partners at risk for HIV. Research suggests that microfinance combined with health promotion can lead to improvement in health outcomes, including reductions in HIV risk and gender-based violence. However, few, if any well designed evaluations of microfinance and health programs with young men have been reported.

ELIGIBILITY:
Inclusion Criteria:

* Must be registered camp member for at least the last 3 months
* Must be at least 15 years old
* Must plan to reside in Dar es Salaam, Tanzania for the next 30 months
* Must visit primary camp at least 1 time per week
* Must provide contact information of friend or family member

Exclusion Criteria:

* Unwilling to provide locator information
* Unable to participate due to psychological disturbance, cognitive impairment or threatening behavior.

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2623 (Actual)
Dates: Start 2013-07; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of New Sexually Transmitted Infections | at 30 months

SECONDARY OUTCOMES:
Proportion of Men Reporting Perpetration of Physical, Sexual, or Psychological Partner Violence | at 12 months
Proportion of Men Reporting Perpetration of Physical, Sexual, or Psychological Partner Violence | at 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Maman, PhD, Principal Investigator — UNC Chapel Hill; Lusajo Kajula-Maonga, MA, Principal Investigator — Muhimbilit University of Health and Allied Sciences
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available on request, and per NIH regulations.

REFERENCES:
- [Background] Kajula L, Balvanz P, Kilonzo MN, Mwikoko G, Yamanis T, Mulawa M, Kajuna D, Hill L, Conserve D, Reyes HL, Leatherman S, Singh B, Maman S. Vijana Vijiweni II: a cluster-randomized trial to evaluate the efficacy of a microfinance and peer health leadership intervention for HIV and intimate partner violence prevention among social networks of young men in Dar es Salaam. BMC Public Health. 2016 Feb 3;16:113. doi: 10.1186/s12889-016-2774-x. PMID 26842360
- [Result] Mulawa M, Kajula LJ, Yamanis TJ, Balvanz P, Kilonzo MN, Maman S. Perpetration and Victimization of Intimate Partner Violence Among Young Men and Women in Dar es Salaam, Tanzania. J Interpers Violence. 2018 Aug;33(16):2486-2511. doi: 10.1177/0886260515625910. Epub 2016 Jan 21. PMID 26802044
- [Result] Mulawa M, Yamanis TJ, Hill LM, Balvanz P, Kajula LJ, Maman S. Evidence of social network influence on multiple HIV risk behaviors and normative beliefs among young Tanzanian men. Soc Sci Med. 2016 Mar;153:35-43. doi: 10.1016/j.socscimed.2016.02.002. Epub 2016 Feb 2. PMID 26874081
- [Result] Mulawa M, Yamanis TJ, Balvanz P, Kajula LJ, Maman S. Comparing Perceptions with Actual Reports of Close Friend's HIV Testing Behavior Among Urban Tanzanian Men. AIDS Behav. 2016 Sep;20(9):2014-22. doi: 10.1007/s10461-016-1335-8. PMID 26880322
- [Result] Hill LM, Maman S, Kilonzo MN, Kajula LJ. Anxiety and depression strongly associated with sexual risk behaviors among networks of young men in Dar es Salaam, Tanzania. AIDS Care. 2017 Feb;29(2):252-258. doi: 10.1080/09540121.2016.1210075. Epub 2016 Jul 28. PMID 27469516
- [Result] Yamanis TJ, Dervisevic E, Mulawa M, Conserve DF, Barrington C, Kajula LJ, Maman S. Social Network Influence on HIV Testing Among Urban Men in Tanzania. AIDS Behav. 2017 Apr;21(4):1171-1182. doi: 10.1007/s10461-016-1513-8. PMID 27506817
- [Result] Mulawa MI, Kajula LJ, Maman S. Peer network influence on intimate partner violence perpetration among urban Tanzanian men. Cult Health Sex. 2018 Apr;20(4):474-488. doi: 10.1080/13691058.2017.1357193. Epub 2017 Aug 16. PMID 28812448
- [Result] Mulawa MI, Reyes HLM, Foshee VA, Halpern CT, Martin SL, Kajula LJ, Maman S. Associations Between Peer Network Gender Norms and the Perpetration of Intimate Partner Violence Among Urban Tanzanian Men: a Multilevel Analysis. Prev Sci. 2018 May;19(4):427-436. doi: 10.1007/s11121-017-0835-8. PMID 28849338